CLINICAL TRIAL: NCT05771701
Title: Pain Pressure Threshold Algometry in Lateral Epicondylitis: Intra- and Inter-rater Reliability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LE1
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Lateral Epicondylitis; Lateral Epicondylitis, Unspecified Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Before starting the investigation, the raters will practice the procedure together in a 30-min training session on a person with lateral epicondylitis. The rater will stabilize the participant's elbow with one hand. The most tender spot in the joint line of each elbow identified by palpation will be assessed with PPT algometry three times with ≥20-second intervals by each rater in a single session. The rubber tip will be placed perpendicular to the skin. The participants will be instructed to give a verbal signal as soon as the sensation of pressure turns into pain, at which time the rater will immediately remove the algometer and record the score. The display of the algometer will face the floor during the testing to blind the raters and participants for the levels of force. There will only be one rater and participant present during the testing at a time. The pause between each rater will be approximately one minute, and the rater order will change randomly during the study period.
Masking Description: The raters will be unaware of each other's test results. Furthermore, the participants will not be informed of their results. Assessor and investigator will be blinded from the providers and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Lateral epicondylitis patients (Experimental): Patients that are diagnosed with lateral epicondylitis.
  Interventions: Device: Pain pressure threshold measurement

INTERVENTIONS:
Device: Pain pressure threshold measurement — Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. The test determines the amount of pressure over a given area in which a steadily increasing nonpainful pressure stimulus turns into a painful pressure sensation. A varying pressure is applied from 0.5 to 1 kg/sec in a perpendicular direction relative to the muscle. PPT has no standard protocol on administration and placement. Equipment used varies with many handheld electric algometers.
  PPT has been used on a wide variety of patients and conditions, including musculoskeletal and neuromuscular disorders (eg, Parkinson disease, tension headaches, pelvic pain, low back pain, myofascial trigger points, sacroiliac joint pain, knee osteoarthritis, skin humidity, shoulder pain, lateral epicondylitis).

SUMMARY:
This clinical trial aims to investigate the intra- and inter-rater reliability of pain pressure threshold algometry in lateral epicondylitis patients.

DETAILED DESCRIPTION:
Tennis elbow, also known as lateral epicondylitis (or epicondylosis) of the elbow, was first described at the end of the 19th century. The community prevalence is 1% to 3%,38 with an even sex distribution and a peak incidence between 35 and 55 years of age.16 There is consensus that the mechanism of injury involves repetitive loads at the wrist and elbow, including supination and extension of the wrist.15 People affected by tennis elbow commonly have pain over the lateral humeral epicondyle, with flexion at the elbow also usually limited by pain, especially if the wrist is pronated and extended against resistance.

Assessment of reliability is a necessary first step in the validation procedures of clinical tests. The reliability of the PPT measurement is susceptible to the influence of rater behavior and judgment, such as the instructions to the participant, rate of force application, and reaction time of the rater.

We opted to investigate the intra- and inter-rater reliability of PPT in persons with lateral epicondylitis with three raters, rater blinding, and a pause of ≥20 seconds between each measurement. We hypothesized that clinicians with no former experience with the procedure can master it with good reliability after a single 30-min training session.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 90 years of age
* Clinical diagnosis of lateral epicondylitis (point tenderness over the lateral epicondyle and exacerbation of pain with chair pick-up test and maximal hand grip)

Exclusion Criteria:

* History of steroid injection for the treatment of lateral epicondylitis within six months
* History of oral steroid use for the treatment of lateral epicondylitis within six months
* History of elbow surgery
* History of elbow fracture
* History of elbow dislocation
* Cancer
* Rheumatoid arthritis
* Severe cognitive deficit
* Neurological deficits in the upper limb
* Inability to speak and understand English/Turkish.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability | 1 day
  Inter-rater reliability of pressure pain threshold measurements using Intraclass Correlation Coefficient (ICC) two-way random model 2.1
Intra-rater reliability | 1 day
  Intra-rater reliability of pressure pain threshold measurements using Intraclass Correlation Coefficient (ICC) two-way random model 2.1

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, Principal Investigator — Uskudar State Hospital
Locations (1):
- Başakşehir Çam ve Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared by the corresponding author upon reasonable request.
Supporting Information: SAP, CSR
Time Frame: 1 year
Access Criteria: Individual participant data will be shared by the corresponding author upon reasonable request.